CLINICAL TRIAL: NCT05459467
Title: Safety and Outcomes of a Structured Exercise Programme in Young Patients With Hypertrophic Cardiomyopathy: the SAFE HCM Trial
Brief Title: Exercise Training in Hypertrophic Cardiomyopathy: (SAFE-HCM)
Acronym: SAFE-HCM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St George's, University of London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 17.0215
Record Dates: First submitted 2020-02-27; First posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Hypertrophic cardiomyopathy; Cardiac rehabilitation; Exercise; High intensity
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Masking for randomisation and analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Participants began exercising at 70% of their heart rate reserve (HRR). The Borg scale was used to monitor exertion during the programme. Participants were provided with watches to monitor their HR and also wore ECG monitors to assess for arrhythmias during exercise classes.
  Sessions consisted of a circuit of set exercises alternating between aerobic/cardiovascular and resistance exercises. Participants were progressed in a graded fashion (up to a maximum of 85% HRR). Participants were also expected to participate in a predefined exercise session remotely.
  Educational session took place in the half an hour following the exercise session. Examples of topics covered included: living with HCM, medications, diet, stress/anxiety management and mindfulness, ICD therapy- what to expect?.
  Interventions: Other: Exercise
- Usual care (No Intervention): Patients exercised as per usual.

INTERVENTIONS:
Other: Exercise — 12 weeks high intensity exercise programme
  Arms: Exercise

SUMMARY:
To explore the feasibility, safety, health and psychological benefits of a 12-week high intensity exercise programme in a young group of individuals with hypertrophic cardiomyopathy (HCM). This will pave the way for a large-scale randomised study of safety of exercise in HCM, the results of which will strengthen the evidence base for exercise recommendations.

DETAILED DESCRIPTION:
A greater understanding of the pathogenic mechanisms underpinning HCM has translated to improved medical care and better survival of affected individuals. Historically these patients were considered to be at high risk of sudden cardiac death during exercise, therefore exercise recommendations were highly conservative and promoted a sedentary life style. There is emerging evidence which suggests that exercise in HCM has a favourable effect on cardiovascular remodelling and moderate exercise programmes have not raised any safety concerns. Furthermore, individuals with HCM have a similar burden of atherosclerotic risk factors as the general population in whom exercise has been associated with a reduction in myocardial infarction, stroke and heart failure, especially among those with a high-risk burden.

Small studies have revealed that athletes who choose to continue with regular competition do not demonstrate adverse outcomes when compared to those who discontinue sport, and active individuals implanted with an implantable cardioverter defibrillator (ICD) do not have an increased risk of appropriate shocks or other adverse events. The recently published exercise recommendations from the European Society of Cardiology account for more contemporary evidence and adopt a more liberal stance regarding competitive and high intensity sport in individuals with low-risk HCM.

However, further work is required into exercise prescription in younger non competitive individuals participating in higher intensity exercise. Moreover low/moderate intensity exercise may be appropriate for older HCM patients, it is unlikely to attract younger, often asymptomatic patients, who wish to engage in higher intensity regimes.Therefore this study aims to assess the feasibility, safety and outcomes of an individually tailored, high intensity exercise programme in young patients with HCM.

ELIGIBILITY:
Inclusion Criteria:

* HCM*
* Age range (16-60 years)
* All genders
* All ethnicities
* Symptomatic and/or asymptomatic HCM patients (NYHA functional class I-II) stable on medication over the preceding 3 months
* Patients may have ICDs
* Patients able to exercise
* Patients able to commit to the full duration of the exercise programme
* Patients able to lie flat

Exclusion Criteria:

* Competitive athletes (individuals who participate in team or individual sports that require systematic training to participate in regular competition against others)
* Exercise induced syncope
* Uncontrolled ventricular arrhythmias (arrhythmias which cause distracting/disabling symptoms or have caused or may cause incapacity)
* NYHA class III-IV
* Severe LV failure (ejection fraction <35%)
* Exercise limited by a non-cardiac (unrelated to HCM) cause
* Surgical myectomy
* Awaiting or recent device implantation (within the last 3 months if due to an arrhythmic events, 4 weeks for primary prevention)
* Known coronary artery disease - defined as a coronary artery lesion of >50% on coronary angiography or known coronary intervention
* Renal failure (eGFR <30ml/min, chronic kidney disease stage 4 and 5 or acute renal failure)
* Patients with Friedrich's ataxia, Noonan syndrome, Anderson-Fabry disease and other disorders associated with cardiac hypertrophy
* Pregnancy

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
Safety composite outcome | 6 months
  This will be reported as the number of people who reach the composite safety outcome (the occurrence of at least one) of the following measured variables 1)cardiovascular death; 2)cardiac arrest; 3) appropriate or inappropriate ICD therapy; 4)exercise induced syncope; 5)sustained ventricular tachycardia; 6) non-sustained ventricular tachycardia; or 7)sustained atrial arrhythmias >30seconds post testing and at 6 months.
Feasibility (qualitative outcome) | 12 weeks
  Feasibility will be reported qualitatively using an open ended questionnaire through analysis of the following a) response to invitation to participate and reasons for refusal; b) adherence to the cardiac rehabilitation programme; c) practical issues related to the programme including staffing and resource assessment; d) acceptability of the intervention and educational materials provided to patients and families

SECONDARY OUTCOMES:
Impact on exercise capacity; time to anaerobic threshold (tAT) (seconds) | 6 months
  This variable will be assessed individually and compared to baseline values post testing and at 6 months.
Impact on exercise capacity; total exercise time (tMax) (seconds) | 6 months
  This variable will be assessed individually and compared to baseline values post testing and at 6 months.
Impact on exercise capacity; VO2(ml/kg/min) at AT (VO2/kgAT) (ml/kg/min) | 6 months
  The anaerobic threshold (AT) was calculated initially using the V slope method (visual estimation from the VCO2 and VO2 graphs at the point where the slope of the VCO2 curve exceeded the slope of the VO2 curve). This was checked manually using the raw data and 10 second averaging. All data was additionally averaged over 10 seconds at this point and the averaged VO2 ml/kg/min value used as the VO2 at the AT. This variable will be assessed individually and compared to baseline values post testing and at 6 months.
Impact on exercise capacity; peak VO2(ml/kg/min) (VO2/kgMax) (ml/kg/min) | 6 months
  CPET analysis was performed using COSMED Quark CPET metabolic cart (Rome, Italy). This automatically calculated peak VO2 ml/min and converted it to ml/kg/min using the patient's weight which had been inputted into the program prior to commencing the CPET. This variable will be assessed individually and compared to baseline values post testing and at 6 months.
Impact on exercise capacity; VE/VCO2 slope (ratio) | 6 months
  This variable will be assessed individually and compared to baseline values post testing and at 6 months.
Impact on exercise capacity; physical activity levels (hours/week) | 6 months
  This variable will be assessed individually and compared to baseline values post testing and at 6 months.
Impact on cardiovascular risk factors; blood pressure (BP) (mmHg) | 6 months
  This variable will be assessed individually and compared to baseline values post testing and at 6 months.
Impact on cardiovascular risk factors; body mass index (BMI) (kg/m2) | 6 months
  This variable will be assessed individually and compared to baseline post testing and at 6 months.
Impact on cardiovascular risk factors; lipid profile (mmol/l) | 12 weeks
  This variable will be assessed individually and compared to baseline values post testing.
Impact on cardiovascular risk factors; HbA1c (mmol/mol) | 12 weeks
  This variable will be assessed individually and compared to baseline values post testing.
Impact on QoL and psychological parameters; Short form 36 (SF36) scores | 6 months
  This variable will be assessed individually and compared to baseline values post testing and at 6 months. The SF-36 is comprised of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is converted into a 0-100 scale, with a lower score denoting greater disability.
Impact on QoL and psychological parameters; Hospital anxiety and depression scale (HADS) scores | 6 months
  This variable will be assessed individually and compared to baseline values post testing and at 6 months. The HADS questionnaire consists of seven items each for depression and anxiety. Each item is scored from zero to three, with three the highest anxiety or depression level. Either an anxiety or depression score of >8 points (total 21) denotes considerable symptoms of anxiety or depression.
Impact on QoL and psychological parameters; WHO disability assessment scale II (WHODAS II) scores | 6 months
  This variable will be assessed individually and compared to baseline values post testing and at 6 months. The WHODAS II score can be calculated using simple scoring where the following scores are assigned to each item - none (1), mild (2) moderate (3), severe (4) and extreme (5). The scores are then summed, with a higher score denoting greater disability.
Impact on disease phenotype-cardiac biomarkers; troponin (ng/l) | 12 weeks
  This variable will be assessed individually and compared to baseline values post testing.
Impact on disease phenotype-cardiac biomarkers; BNP (ng/l) | 12 weeks
  This variable will be assessed individually and compared to baseline values post testing.
Impact on disease phenotype-echocardiographic outcomes; LA volume (ml) | 12 weeks
  This variable will be assessed individually and compared to baseline values post testing.
Impact on disease phenotype-echocardiographic outcomes; LVEDD (mm) | 12 weeks
  This variable will be assessed individually and compared to baseline values post testing.
Impact on disease phenotype-echocardiographic outcomes; LVWT (mm) | 12 weeks
  This variable will be assessed individually and compared to baseline values post testing.
Impact on disease phenotype-echocardiographic outcomes; diastolic parameters (E/E', E/A)) | 12 weeks
  This variable will be assessed individually and compared to baseline values post testing.
Impact on disease phenotype-ventricular ectopic burden; | 6 months
  The absolute number of ventricular ectopics will be assessed and compared to baseline values post testing post testing and at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Papadakis, Principal Investigator — St George's University London
Locations (3):
- United Kingdom (3):
  - Guys and St Thomas's Hospital, London
  - Kings College Hospital, London
  - St George's Hospital, London

IPD SHARING:
Plan to Share IPD: No
Currently individual participant data will not be shared with other researchers.